CLINICAL TRIAL: NCT02830334
Title: Use of the Ask Suicide-Screening Questions (ASQ) in Pediatric Outpatient Settings
Status: Terminated | Type: Observational
Why Stopped: this study was determined by IRB not to be humans subjects research
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999916130; 16-M-N130
Record Dates: First submitted 2016-07-09; First posted 2016-07-12 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Adolescents; Children
Keywords: Suicide; Youth Suicide
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

Doctors and nurses who work in non-mental health settings need ways to know when patients are at risk. Researchers created the Ask Suicide-Screening Questions (ASQ) to be used in an emergency department for children. This is a 4-item suicide risk screening tool. We wanted to see if this is also a good tool to use in the outpatient setting. Two studies are being done to test it at hospitals. This study is for researchers to analyze the data from those two studies.

Objectives:

To combine and analyze data from two studies to see how well the ASQ can detect suicide risk in pediatric outpatient clinics.

Eligibility:

No people are enrolled in this study.

Design:

Participants in the two non-NIH studies will give consent for their data to be shared.

The data will be confidential and secure. They will have no personal information attached to them.

Researchers will get the data and analyze them.

DETAILED DESCRIPTION:
This protocol is designed to combine and analyze data from two separate independent studies conducted at non-NIH sites-Boston Children s Hospital (BCH) and Kansas City Mercy Children s Hospital (KC). Both sites have protocols and consents reviewed by the IRBs at their respective institutions, and data collection is underway; NIMH will coordinate and oversee data analysis from these studies. A protocol to establish NIH s role in the studies and IRB review will enhance the acceptance of the research findings for publication in scientific and medical journals.

Physicians and nurses working in non-mental health settings require tools to guide them in recognizing patients at risk. While screening children and adolescents is emerging as a priority of the Joint Commission, there are currently no suicide screening instruments designed specifically for assessing suicide risk in a pediatric outpatient medical setting. Recently, our study team developed the Ask Suicide-Screening Questions (ASQ), a 4-item suicide risk screening instrument with excellent sensitivity, specificity, and negative predictive value for use in pediatric emergency departments (Protocol 08-M-N070). However, use of the ASQ in an outpatient medical setting has not been tested. The aim of the studies at BCH and KC is to determine the utility of the ASQ among youth in outpatient primary and specialty care clinics (e.g., endocrine, sports medicine, orthopedic). While most outpatients will not be at imminent risk for suicide, we hypothesize that the ASQ will capture a number of patients who screen positive and are not only at risk for suicidal behavior in the future, but are also experiencing significant emotional distress and therefore warrant further psychiatric evaluation and follow-up treatment. Data from BCH and KC will be analyzed under this protocol from a total sample size of 580. Two measures of suicide risk (the ASQ and the Suicidal Ideation Questionnaire) and a depression screen (the Patient Health Questionnaire - Adolescent version), are administered to all eligible patients aged 10-21 years. The ultimate goal is to provide non-mental health clinicians with a brief, accurate assessment tool for detecting risk of suicide in pediatric medical outpatients and in turn, connecting those in need with mental health services.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patient in the Adolescent/Young Adult Medicine Program.
* English-speaking
* Aged 10-21 years, inclusive.
* If 18 or older, can supply consent.
* If under 18, has a parent or legal guardian who is available for informed consent (written/verbal).

EXCLUSION CRITERIA:

* Has a severe developmental or cognitive delay.
* Has a severe communication disorder such that the patient cannot comprehend questions or communicate answers.
* Has a severe illness that prevents adequate communication.
* Parents/guardians and/or patients are non-English speaking.
* Patients under 18 years old are not with a parent/legal guardian who can provide written consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 525 (Actual)
Dates: Start 2016-07-09 (Actual); Primary Completion 2018-05-10 (Actual); Study Completion 2020-04-22 (Actual)

PRIMARY OUTCOMES:
Primary outcome measures include frequencies of positive responses to all ASQ and SIQ items. | Ongoing

SECONDARY OUTCOMES:
Responses to demographic survey items will allow us to describe if the primary outcome measure varies by race, gender, education level, and other demographic variables. A depression screen and a brief questionnaire to assess parent opinion will... | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Horowitz, Ph.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (2):
- United States (2):
  - Childrens Hospital, Boston, Boston, Massachusetts
  - The Childrens Mercy Hospital, Kansas City, Missouri